CLINICAL TRIAL: NCT00143663
Title: A Double-blind, Randomized Study to Evaluate the Efficacy and Safety of TAK-475 100 mg Versus Placebo in Subjects With Primary Hypercholesterolemia
Brief Title: Effect of Lapaquistat Acetate on Blood Cholesterol Levels in Subjects With Elevated Cholesterol
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-475-008; U1111-1122-7722 (Registry Identifier: WHO)
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Dyslipidemia
Keywords: Hypercholesterolemia; Hyperlipidemia; Drug Therapy
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 100 mg QD (Experimental)
  Interventions: Drug: Lapaquistat Acetate
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lapaquistat Acetate — Lapaquistat acetate 100 mg, tablets, orally, once daily for up to 12 weeks
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD
Drug: Placebo — Lapaquistat acetate placebo-matching tablets, orally, once daily for up to 12 weeks
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine if patients with elevated cholesterol, but not taking any other lipid medication, could lower their cholesterol with administration of lapaquistat acetate, once daily (QD).

DETAILED DESCRIPTION:
This study will evaluate the efficacy and safety of TAK-475 (lapaquistat acetate) compared to placebo in subjects with primary hypercholesterolemia. Subjects who have signed the informed consent will undergo necessary evaluations to determine eligibility for a dietary run-in phase. Subjects who meet randomization criteria will enter treatment with one of the following randomized treatments: lapaquistat acetate or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of childbearing potential cannot be been pregnant, lactating and are not planning on becoming pregnant and agrees to use acceptable forms of contraception throughout the course of this study.
* Must have a mean low-density lipoprotein cholesterol values between 3.367 and 5.689 mmol/L, inclusive, from 2 consecutive samples taken at least 1 week apart with the difference between the 2 values not exceeding 15% of the higher value.
* Must have a triglyceride value of 4.516 mmol/L or less from 2 consecutive samples taken at least 1 week apart with the upper value from either sample being 5.081 mmol/L or less.
* Has clinical laboratory evaluations within the reference ranges for the testing laboratory unless the results were deemed not clinically significant by the investigator or sponsor.
* Is willing and able to maintain a standardized low-cholesterol diet.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level greater than 1.5 times the upper limit of normal, active liver disease or jaundice.
* Has a serum creatinine level greater than 135 μmol/L.
* Has a creatine phosphokinase value greater than three times the upper limit of normal.
* Has diabetes mellitus type 1 or 2.
* Has a history of cancer that had been in remission for less than 5 years prior to the first dose of study drug. This criterion did not include subjects with basal cell or stage I squamous cell carcinoma of the skin.
* Has an endocrine disorder, such as Cushing syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a history of myocardial infarction, angina pectoris, transient ischemic attacks, cerebrovascular accident, peripheral vascular disease, abdominal aortic aneurysm, coronary revascularization or multiple risk factors that present a 10-year risk for CHD of greater than 20%, based on Framingham risk scoring.
* Has a positive hepatitis B surface antigen or hepatitis C virus antibody, as determined by medical history and/or participant's verbal report.
* Has a positive human immunodeficiency virus test result or was taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Is unable or unwilling to discontinue excluded medications or to continue stable doses of "stable dose" medications or would require treatment with any excluded medication during the study.
* Has had exposure to lapaquistat acetate in other studies or was participating or enrolled in another investigational study within the previous 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's half-life.
* Has a history or presence of a clinically significant food allergy that would prevent adherence to the therapeutic lifestyle change (or equivalent) diet.
* Has a known heterozygous or homozygous familial hypercholesterolemia or known type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension.
* Has inflammatory bowel disease or any other malabsorption syndrome or had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or alcohol abuse within the past 2 years.
* Has any other serious disease or condition at Run-In or at Randomization that might reduce life expectancy, impair successful management according to the protocol, or make the subject an unsuitable candidate to receive study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2005-09; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Low-Density Lipoprotein cholesterol | Week 12 or Final Visit

SECONDARY OUTCOMES:
Change from Baseline in Calculated Low-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in High-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Low-Density Lipoprotein cholesterol/ High-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Very Low-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in non- High-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in Triglycerides | Week 12 or Final Visit
Change from Baseline in Total Cholesterol | Week 12 or Final Visit
Change from Baseline in the ratio of Total Cholesterol/High-Density Lipoprotein cholesterol | Week 12 or Final Visit
Change from Baseline in apolipoprotein A1 | Week 12 or Final Visit
Change from Baseline in apolipoprotein B | Week 12 or Final Visit
Change from Baseline in the ratio of apolipoprotein B/ apolipoprotein A1 | Week 12 or Final Visit
Change from Baseline in High-Sensitivity C-reactive Protein | Week 12 or Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (47):
- United States (47):
  - Northport, Alabama
  - Mesa, Arizona
  - Chula Vista, California
  - Encinitas, California
  - Long Beach, California
  - Pismo Beach, California
  - Sacramento, California
  - San Diego, California
  - Golden, Colorado
  - Aventura, Florida
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - New Port Richy, Florida
  - Pembroke Pines, Florida
  - Elk Grove Village, Illinois
  - Peoria, Illinois
  - Evansville, Indiana
  - Indianapolis, Indiana
  - Arkansas City, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Livonia, Michigan
  - Las Vegas, Nevada
  - Margate City, New Jersey
  - New Hyde Park, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Statesville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Medford, Oregon
  - Downingtown, Pennsylvania
  - Sellersville, Pennsylvania
  - Tipton, Pennsylvania
  - Warwick, Rhode Island
  - Charleston, South Carolina
  - Mt. Pleasant, South Carolina
  - Bristol, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Norfolk, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985